CLINICAL TRIAL: NCT02607865
Title: Efficacy and Long-term Safety of Oral Semaglutide Versus Sitagliptin in Subjects With Type 2 Diabetes
Acronym: PIONEER 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-4222; 2015-001351-71 (EudraCT Number); U1111-1168-4339 (Other: WHO); JAPIC (Other: JapicCTI-163174)
Record Dates: First submitted 2015-11-10; First posted 2015-11-18 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Semaglutide 3 mg (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- Semaglutide 7 mg (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- Semaglutide 14 mg (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- Sitagliptin 100 mg (Active Comparator)
  Interventions: Drug: sitagliptin; Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Oral administration once-daily
  Arms: Semaglutide 14 mg; Semaglutide 3 mg; Semaglutide 7 mg
Drug: sitagliptin — Oral administration once-daily
  Arms: Sitagliptin 100 mg
Drug: placebo — Oral administration once-daily

SUMMARY:
This trial is conducted globally. The aim of the trial is to investigate efficacy and long-term safety of oral semaglutide versus sitagliptin in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at least 18 years at the time of signing informed consent For Japan only: Male or female, age at least 20 years at the time of signing informed consent
* Diagnosed with T2DM (type 2 diabetes mellitus) for at least 90 days prior to day of screening
* HbA1c (glycosylated haemoglobin) 7.0-10.5 % (53-91 mmol/mol) (both inclusive).
* Stable daily dose of metformin (equal or above 1500 mg or maximum tolerated dose as documented in subject medical record) alone or in combination with SU (= half of the maximum approved dose according to local label or maximum tolerated dose as documented in subject medical record) within 90 days prior to the day of screening

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice). For certain specific countries: Additional specific requirements apply
* Family or personal history of Multiple Endocrine Neoplasia Type 2 (MEN 2) or Medullary Thyroid Carcinoma (MTC)
* History of pancreatitis (acute or chronic)
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* Any of the following: myocardial infarction, stroke or hospitalization for unstable angina and/or transient ischaemic attack within the past 180 days prior to the day of screening
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV.
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening.
* Renal impairment defined as estimated Glomerular Filtration Rate (eGFR) below 60 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and in-situ carcinomas)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1864 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (205):
- United States (84):
  - Novo Nordisk Investigational Site, Anniston, Alabama
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Tuscumbia, Alabama
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Carmichael, California
  - Novo Nordisk Investigational Site, Coronado, California
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Los Alamitos, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Port Charlotte, Florida
  - Novo Nordisk Investigational Site, Spring Hill, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Perry, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Park City, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Natchitoches, Louisiana
  - Novo Nordisk Investigational Site, Shreveport, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Flint, Michigan
  - Novo Nordisk Investigational Site, Sterling Heights, Michigan
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Teaneck, New Jersey
  - Novo Nordisk Investigational Site, Trenton, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, High Point, North Carolina
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Maumee, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, Corvallis, Oregon
  - Novo Nordisk Investigational Site, Jersey Shore, Pennsylvania
  - Novo Nordisk Investigational Site, McMurray, Pennsylvania
  - Novo Nordisk Investigational Site, Gaffney, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Pelzer, South Carolina
  - Novo Nordisk Investigational Site, Summerville, South Carolina
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Jackson, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Longview, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Waco, Texas
  - Novo Nordisk Investigational Site, Murray, Utah
  - Novo Nordisk Investigational Site, South Burlington, Vermont
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Argentina (3):
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Córdoba
- Novo Nordisk Investigational Site, São Paulo, São Paulo, Brazil
- France (15):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Châlons-en-Champagne
  - Novo Nordisk Investigational Site, Dijon
  - Novo Nordisk Investigational Site, La Roche-sur-Yon
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Limoges
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Perpignan
  - Novo Nordisk Investigational Site, Périgueux
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (12):
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Elsterwerda
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Stuttgart
- India (12):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Gurgaon, Haryana
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Bhubaneshwar, Odisha
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
- Israel (7):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Raanana
  - Novo Nordisk Investigational Site, Tel Aviv
- Japan (13):
  - Novo Nordisk Investigational Site, Asahikawa-shi, Hokkaido
  - Novo Nordisk Investigational Site, Gunma
  - Novo Nordisk Investigational Site, Hokkaido
  - Novo Nordisk Investigational Site, Ibaraki
  - Novo Nordisk Investigational Site, Iruma-shi, Saitama
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Kyoto-shi, Kyoto
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Shizuoka-shi, Shizuoka
  - Novo Nordisk Investigational Site, Tokyo
- Mexico (5):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Toluca, State of Mexico
  - Novo Nordisk Investigational Site, Ciudad Madero, Tamaulipas
  - Novo Nordisk Investigational Site, Aguascalientes
  - Novo Nordisk Investigational Site, San Luis Potosí City
- Romania (11):
  - Novo Nordisk Investigational Site, Piteşti, Argeş
  - Novo Nordisk Investigational Site, Oradea, Bihor County
  - Novo Nordisk Investigational Site, Craiova, Dolj
  - Novo Nordisk Investigational Site, Baia Mare, Maramureş
  - Novo Nordisk Investigational Site, Târgu Mureş, Mureș County
  - Novo Nordisk Investigational Site, Ploieşti, Prahova
  - Novo Nordisk Investigational Site, Timișoara, Timiș County
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Iași
  - Novo Nordisk Investigational Site, Satu Mare
  - Novo Nordisk Investigational Site, Timișoara
- Russia (6):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Yaroslavl
- South Africa (9):
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Krugersdorp, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
  - Novo Nordisk Investigational Site, Cape Town
  - Novo Nordisk Investigational Site, Pretoria
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
  - Novo Nordisk Investigational Site, Samsun
- Ukraine (8):
  - Novo Nordisk Investigational Site, Cherkasy
  - Novo Nordisk Investigational Site, Ivano-Frankivsk
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Mykolaiv
  - Novo Nordisk Investigational Site, Odesa
  - Novo Nordisk Investigational Site, Ternopil
  - Novo Nordisk Investigational Site, Zaporizhia
  - Novo Nordisk Investigational Site, Zhytomyr
- United Kingdom (15):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, Chester
  - Novo Nordisk Investigational Site, Crewe
  - Novo Nordisk Investigational Site, Doncaster
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Preston
  - Novo Nordisk Investigational Site, Rotherham
  - Novo Nordisk Investigational Site, Sidcup
  - Novo Nordisk Investigational Site, Soham
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Taunton
  - Novo Nordisk Investigational Site, Torquay
  - Novo Nordisk Investigational Site, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Rosenstock J, Allison D, Birkenfeld AL, Blicher TM, Deenadayalan S, Jacobsen JB, Serusclat P, Violante R, Watada H, Davies M; PIONEER 3 Investigators. Effect of Additional Oral Semaglutide vs Sitagliptin on Glycated Hemoglobin in Adults With Type 2 Diabetes Uncontrolled With Metformin Alone or With Sulfonylurea: The PIONEER 3 Randomized Clinical Trial. JAMA. 2019 Apr 16;321(15):1466-1480. doi: 10.1001/jama.2019.2942. PMID 30903796
- [Result] Araki E, Terauchi Y, Watada H, Deenadayalan S, Christiansen E, Horio H, Kadowaki T. Efficacy and safety of oral semaglutide in Japanese patients with type 2 diabetes: A post hoc subgroup analysis of the PIONEER 1, 3, 4 and 8 trials. Diabetes Obes Metab. 2021 Dec;23(12):2785-2794. doi: 10.1111/dom.14536. Epub 2021 Sep 27. PMID 34472698
- [Result] Eliasson B, Ericsson A, Fridhammar A, Nilsson A, Persson S, Chubb B. Long-Term Cost Effectiveness of Oral Semaglutide Versus Empagliflozin and Sitagliptin for the Treatment of Type 2 Diabetes in the Swedish Setting. Pharmacoecon Open. 2022 May;6(3):343-354. doi: 10.1007/s41669-021-00317-z. Epub 2022 Jan 21. PMID 35064550
- [Result] Aroda VR, Bauer R, Christiansen E, Haluzik M, Kallenbach K, Montanya E, Rosenstock J, Meier JJ. Efficacy and safety of oral semaglutide by subgroups of patient characteristics in the PIONEER phase 3 programme. Diabetes Obes Metab. 2022 Jul;24(7):1338-1350. doi: 10.1111/dom.14710. Epub 2022 May 9. PMID 35373893
- [Derived] Pulleyblank R, Larsen NB. Cost-Effectiveness of Semaglutide vs. Empagliflozin, Canagliflozin, and Sitagliptin for Treatment of Patients with Type 2 Diabetes in Denmark: A Decision-Analytic Modelling Study. Pharmacoecon Open. 2023 Jul;7(4):579-591. doi: 10.1007/s41669-023-00416-z. Epub 2023 May 13. PMID 37178435
- [Derived] Pratley RE, Crowley MJ, Gislum M, Hertz CL, Jensen TB, Khunti K, Mosenzon O, Buse JB. Oral Semaglutide Reduces HbA1c and Body Weight in Patients with Type 2 Diabetes Regardless of Background Glucose-Lowering Medication: PIONEER Subgroup Analyses. Diabetes Ther. 2021 Apr;12(4):1099-1116. doi: 10.1007/s13300-020-00994-9. Epub 2021 Mar 4. PMID 33660198
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Thethi TK, Pratley R, Meier JJ. Efficacy, safety and cardiovascular outcomes of once-daily oral semaglutide in patients with type 2 diabetes: The PIONEER programme. Diabetes Obes Metab. 2020 Aug;22(8):1263-1277. doi: 10.1111/dom.14054. Epub 2020 May 13. PMID 32267058
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 200 sites in 14 countries: Argentina-5, Brazil-1, France-10, Germany-12, Israel-8, Japan-16, Mexico-5, Romania-12, Russian Federation-8, South Africa-11, Turkey-7, Ukraine-8, United Kingdom (UK)-14, United States (US)-83. In addition, 6 sites screened, but didn't randomise any subjects: France-1, Turkey-1, UK-1 and US-3.
Pre-assignment Details: Data presented in "participant flow" is based on the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide 3 mg: Participants were to take oral semaglutide 3 mg tablets once daily from week 0 to week 78. In addition, participants were to take sitagliptin placebo tablets once daily from week 0 to week 78.
- Oral Semaglutide 7 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 78: 3 mg from week 0 to week 4 and 7 mg from week 4 to week 78. In addition, participants were to take sitagliptin placebo tablets once daily from week 0 to week 78.
- Oral Semaglutide 14 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 78: 3 mg from week 0 to week 4, 7 mg from week 4 to week 8 and 14 mg from week 8 to week 78. In addition, participants were to take sitagliptin placebo tablets once daily from week 0 to week 78.
- Sitagliptin 100 mg: Participants were to take sitagliptin 100 mg tablets once daily from week 0 to week 78. In addition, participants were to take oral semaglutide placebo tablets once daily from week 0 to week 78.
Period: Overall Study
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Started | 466 | 466 | 465 | 467
Full Analysis Set (FAS) (One participant was excluded from the FAS as the participant was a confirmed screening failure.) | 466 | 465 | 465 | 467
Safety Analysis Set (SAS) | 466 | 464 | 465 | 466
Completed | 433 | 436 | 438 | 451
Not Completed | 33 | 30 | 27 | 16
Not completed — Lost to Follow-up | 9 | 7 | 7 | 5
Not completed — Withdrawal by Subject | 18 | 18 | 17 | 8
Not completed — Death | 5 | 4 | 1 | 3
Not completed — Unclassified | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The FAS comprised all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg | Total
Number analyzed (Participants) | 466 | 465 | 465 | 467 | 1863
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10) | 58 (10) | 57 (10) | 58 (10) | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 220 | 218 | 229 | 879
  Male | 254 | 245 | 247 | 238 | 984
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was recorded as 'Not Applicable' for Brazil and France.
  Participants
    White | 344 | 330 | 317 | 333 | 1324
    Black or African American | 38 | 38 | 45 | 39 | 160
    Asian | 56 | 69 | 61 | 59 | 245
    American Indian or Alaska Native | 4 | 3 | 5 | 6 | 18
    Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 1
    Other | 13 | 11 | 20 | 12 | 56
    Not applicable | 10 | 14 | 17 | 18 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity was recorded as 'Not Applicable' for France.
  Participants
    Hispanic or Latino | 76 | 77 | 75 | 93 | 321
    Not Hispanic or Latino | 385 | 378 | 377 | 366 | 1506
    Not applicable | 5 | 10 | 13 | 8 | 36
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.3 (1.0) | 8.4 (1.0) | 8.3 (0.9) | 8.3 (0.9) | 8.3 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c: Week 26
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated at week 26. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. The endpoint was also evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Percentage of HbA1c
  In-trial: number analyzed (Participants) | 435 | 438 | 436 | 446
  In-trial | -0.6 (1.0) | -1.1 (1.1) | -1.3 (1.0) | -0.8 (0.9)
  On-treatment without rescue medication: number analyzed (Participants) | 391 | 409 | 398 | 419
  On-treatment without rescue medication | -0.6 (1.0) | -1.2 (1.1) | -1.4 (1.0) | -0.8 (0.9)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Sitagliptin 100 mg; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an analysis of covariance (ANCOVA) model with treatment, strata, and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Non-Inferiority — This hypothesis was controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand). A value of 0.3% (the non-inferiority margin) was added to imputed values at week 26 for the oral semaglutide treatment arm only; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from the non-inferiority margin (non-inferiority). The non-inferiority margin was 0.3%; Mean treatment difference = -0.5, 95% CI 2-sided [-0.6 to -0.4] — Oral semaglutide 14 mg - Sitagliptin 100 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 14 mg vs Sitagliptin 100 mg; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an ANCOVA model with treatment, strata, and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — This hypothesis was controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand); p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.5, 95% CI 2-sided [-0.6 to -0.4] — Oral semaglutide 14 mg - Sitagliptin 100 mg
Statistical Analysis 3: Comparison: Oral Semaglutide 7 mg vs Sitagliptin 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Pattern mixture model — [p-value comment as in outcome 1, analysis 1]; Mean treatment difference = -0.2, 95% CI 2-sided [-0.4 to -0.1] — Oral semaglutide 7 mg - Sitagliptin 100 mg
Statistical Analysis 4: Comparison: Oral Semaglutide 7 mg vs Sitagliptin 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.3, 95% CI 2-sided [-0.4 to -0.1] — Oral semaglutide 7 mg - Sitagliptin 100 mg
Statistical Analysis 5: Comparison: Oral Semaglutide 3 mg vs Sitagliptin 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0856, Pattern mixture model — [p-value comment as in outcome 1, analysis 1]; Mean treatment difference = 0.2, 95% CI 2-sided [0.1 to 0.3] — Oral semaglutide 3 mg - Sitagliptin 100 mg
Statistical Analysis 6: Comparison: Oral Semaglutide 3 mg vs Sitagliptin 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — This hypothesis was not controlled for multiplicity, since the non-inferiority test of change in HbA1c for oral semaglutide 3 mg versus sitagliptin 100 mg could not be confirmed. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand); p = 0.0080, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = 0.2, 95% CI 2-sided [0.0 to 0.3] — Oral semaglutide 3 mg - Sitagliptin 100 mg. If the mean treatment difference is non-negative, the superiority hypothesis of oral semaglutide 3 mg vs sitagliptin 100 mg will never be confirmed irrespective of the observed two-sided p-value
Statistical Analysis 7: Comparison: Oral Semaglutide 14 mg vs Sitagliptin 100 mg; The analysis was based on a mixed model for repeated measurements (MMRM) that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment, strata and region as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Non-Inferiority — This hypothesis was not controlled for multiplicity. Results are based on the data from the on-treatment without rescue medication observation period. The estimated treatment effect excludes the effect of any rescue medication and any effect after premature trial product discontinuation (hypothetical estimand); p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Mean treatment difference = -0.6, 95% CI 2-sided [-0.7 to -0.5] — Oral semaglutide 14 mg - Sitagliptin 100 mg
Statistical Analysis 8: Comparison: Oral Semaglutide 14 mg vs Sitagliptin 100 mg; The analysis was based on a MMRM that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment, strata and region as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.6, 95% CI 2-sided [-0.7 to -0.5] — Oral semaglutide 14 mg - Sitagliptin 100 mg
Statistical Analysis 9: Comparison: Oral Semaglutide 7 mg vs Sitagliptin 100 mg; [analysis description as in outcome 1, analysis 8]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 7]; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Mean treatment difference = -0.3, 95% CI 2-sided [-0.4 to -0.2] — Oral semaglutide 7 mg - Sitagliptin 100 mg
Statistical Analysis 10: Comparison: Oral Semaglutide 7 mg vs Sitagliptin 100 mg; [analysis description as in outcome 1, analysis 8]; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.3, 95% CI 2-sided [-0.4 to -0.2] — Oral semaglutide 7 mg - Sitagliptin 100 mg
Statistical Analysis 11: Comparison: Oral Semaglutide 3 mg vs Sitagliptin 100 mg; [analysis description as in outcome 1, analysis 8]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 7]; p = 0.3851, MMRM — [p-value comment as in outcome 1, analysis 1]; Mean treatment difference = 0.2, 95% CI 2-sided [0.1 to 0.4] — Oral semaglutide 3 mg - Sitagliptin 100 mg
Statistical Analysis 12: Comparison: Oral Semaglutide 3 mg vs Sitagliptin 100 mg; [analysis description as in outcome 1, analysis 8]; Test type: Other — [test comment as in outcome 1, analysis 7]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = 0.2, 95% CI 2-sided [0.1 to 0.4] — [estimate comment as in outcome 1, analysis 6]

2. Secondary Outcome: Change in Body Weight: Week 26
Description: Change from baseline (week 0) in body weight was evaluated at week 26. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. The endpoint was also evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Kg
  In-trial: number analyzed (Participants) | 438 | 440 | 439 | 447
  In-trial | -1.2 (3.2) | -2.2 (3.9) | -3.1 (3.8) | -0.6 (3.2)
  on-treatment without rescue medication: number analyzed (Participants) | 394 | 411 | 401 | 420
  on-treatment without rescue medication | -1.2 (3.3) | -2.2 (4.0) | -3.2 (3.8) | -0.6 (3.2)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Sitagliptin 100 mg; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an ANCOVA model with treatment, strata, and region as categorical fixed effects and baseline body weight value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -2.5, 95% CI 2-sided [-3.0 to -2.0] — Oral semaglutide 14 mg - Sitagliptin 100 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -1.6, 95% CI 2-sided [-2.0 to -1.1] — Oral semaglutide 7 mg - Sitagliptin 100 mg
Statistical Analysis 3: Comparison: Oral Semaglutide 3 mg vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 6]; p = 0.0185, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.6, 95% CI 2-sided [-1.1 to -0.1] — Oral semaglutide 3 mg - Sitagliptin 100 mg
Statistical Analysis 4: Comparison: Oral Semaglutide 14 mg vs Sitagliptin 100 mg; The analysis was based on a MMRM that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment, strata and region as categorical fixed effects and the baseline body weight value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -2.6, 95% CI 2-sided [-3.1 to -2.1] — Oral semaglutide 14 mg - Sitagliptin 100 mg
Statistical Analysis 5: Comparison: Oral Semaglutide 7 mg vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -1.5, 95% CI 2-sided [-2.0 to -1.1] — Oral semaglutide 7 mg - Sitagliptin 100 mg
Statistical Analysis 6: Comparison: Oral Semaglutide 3 mg vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p = 0.0257, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); type Mean treatment difference = -0.5, 95% CI 2-sided [-1.0 to -0.1] — Oral semaglutide 3 mg - Sitagliptin 100 mg

3. Secondary Outcome: Change in HbA1c: Weeks 52 and 78
Description: Change from baseline (week 0) in HbA1c was evaluated at weeks 52 and 78. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Percentage of HbA1c
  Week 52: number analyzed (Participants) | 427 | 431 | 434 | 436
  Week 52 | -0.6 (1.1) | -1.0 (1.2) | -1.2 (1.1) | -0.7 (1.1)
  Week 78: number analyzed (Participants) | 421 | 424 | 425 | 439
  Week 78 | -0.6 (1.1) | -0.9 (1.3) | -1.1 (1.1) | -0.7 (1.1)

4. Secondary Outcome: Change in Body Weight (kg): Weeks 52 and 78
Description: Change from baseline (week 0) in body weight was evaluated at weeks 52 and 78. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Kg
  Week 52: number analyzed (Participants) | 428 | 433 | 435 | 437
  Week 52 | -1.6 (4.1) | -2.5 (4.9) | -3.5 (4.7) | -0.7 (3.7)
  Week 78: number analyzed (Participants) | 425 | 425 | 428 | 443
  Week 78 | -1.8 (4.9) | -2.8 (5.4) | -3.2 (4.9) | -1.0 (4.1)

5. Secondary Outcome: Change in Body Weight (%)
Description: Relative change from baseline (week 0) in body weight (kg) was evaluated at weeks 26, 52 and 78. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Percentage change
  Week 26: number analyzed (Participants) | 438 | 440 | 439 | 447
  Week 26 | -1.23 (3.57) | -2.36 (4.09) | -3.44 (4.21) | -0.64 (3.38)
  Week 52: number analyzed (Participants) | 428 | 433 | 435 | 437
  Week 52 | -1.65 (4.28) | -2.63 (5.09) | -3.83 (5.14) | -0.76 (3.91)
  Week 78: number analyzed (Participants) | 425 | 425 | 428 | 443
  Week 78 | -1.87 (4.87) | -2.92 (5.67) | -3.47 (5.34) | -0.99 (4.39)

6. Secondary Outcome: Change in FPG
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated at weeks 26, 52 and 78. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
mmol/L
  Week 26: number analyzed (Participants) | 433 | 436 | 433 | 443
  Week 26 | -0.83 (2.69) | -1.17 (2.54) | -1.67 (2.60) | -0.90 (2.32)
  Week 52: number analyzed (Participants) | 419 | 429 | 432 | 433
  Week 52 | -0.98 (2.78) | -1.28 (2.62) | -1.75 (2.57) | -1.03 (2.60)
  Week 78: number analyzed (Participants) | 418 | 419 | 419 | 434
  Week 78 | -1.07 (3.21) | -1.11 (2.92) | -1.65 (2.71) | -0.91 (2.59)

7. Secondary Outcome: Change in BMI
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at weeks 26, 52 and 78. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Kg/m^2
  Week 26: number analyzed (Participants) | 438 | 440 | 439 | 447
  Week 26 | -0.4 (1.2) | -0.8 (1.4) | -1.1 (1.4) | -0.2 (1.1)
  Week 52: number analyzed (Participants) | 428 | 433 | 435 | 437
  Week 52 | -0.6 (1.5) | -0.9 (1.7) | -1.2 (1.7) | -0.3 (1.3)
  Week 78: number analyzed (Participants) | 425 | 425 | 428 | 443
  Week 78 | -0.7 (1.8) | -1.0 (1.9) | -1.1 (1.7) | -0.4 (1.5)

8. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated at weeks 26, 52 and 78. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
cm
  Week 26: number analyzed (Participants) | 438 | 439 | 438 | 445
  Week 26 | -0.7 (5.0) | -1.8 (5.2) | -2.3 (5.2) | -0.6 (4.4)
  Week 52: number analyzed (Participants) | 426 | 432 | 435 | 436
  Week 52 | -1.3 (5.7) | -2.3 (6.8) | -2.6 (6.2) | -0.5 (5.1)
  Week 78: number analyzed (Participants) | 424 | 424 | 428 | 440
  Week 78 | -1.2 (6.0) | -2.4 (7.2) | -2.4 (6.1) | -0.7 (5.6)

9. Secondary Outcome: Change in Total Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in total cholesterol (mmol/L) at weeks 26, 52 and 78 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Ratio of total cholesterol
  Week 26: number analyzed (Participants) | 433 | 437 | 432 | 444
  Week 26 | 1.00 (16.8) | 0.98 (17.5) | 0.97 (17.1) | 1.00 (16.4)
  Week 52: number analyzed (Participants) | 421 | 427 | 432 | 435
  Week 52 | 1.00 (17.5) | 0.99 (18.5) | 0.98 (17.0) | 1.01 (16.9)
  Week 78: number analyzed (Participants) | 419 | 419 | 421 | 438
  Week 78 | 1.00 (18.3) | 0.99 (19.3) | 0.99 (18.7) | 1.00 (19.4)

10. Secondary Outcome: Change in LDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in low-density lipoprotein (LDL) cholesterol (mmol/L) at weeks 26, 52 and 78 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Ratio of LDL cholesterol
  Week 26: number analyzed (Participants) | 433 | 437 | 431 | 444
  Week 26 | 1.02 (28.2) | 0.98 (28.0) | 0.98 (28.6) | 1.02 (26.4)
  Week 52: number analyzed (Participants) | 421 | 427 | 431 | 435
  Week 52 | 1.02 (28.1) | 0.99 (29.7) | 0.99 (27.4) | 1.03 (27.7)
  Week 78: number analyzed (Participants) | 419 | 419 | 420 | 438
  Week 78 | 1.03 (30.8) | 1.00 (30.2) | 1.00 (30.2) | 1.03 (32.6)

11. Secondary Outcome: Change in VLDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in very-low-density lipoprotein (VLDL) cholesterol (mmol/L) at weeks 26, 52 and 78 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Ratio of VLDL cholesterol
  Week 26: number analyzed (Participants) | 433 | 437 | 431 | 444
  Week 26 | 0.99 (36.4) | 0.96 (36.1) | 0.91 (36.3) | 0.97 (34.1)
  Week 52: number analyzed (Participants) | 421 | 427 | 431 | 435
  Week 52 | 1.00 (35.0) | 0.98 (39.1) | 0.93 (39.6) | 0.98 (34.4)
  Week 78: number analyzed (Participants) | 419 | 419 | 420 | 438
  Week 78 | 0.95 (41.7) | 0.94 (41.5) | 0.91 (40.4) | 0.94 (39.6)

12. Secondary Outcome: Change in HDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in high-density lipoprotein (HDL) cholesterol (mmol/L) at weeks 26, 52 and 78 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Ratio of HDL cholesterol
  Week 26: number analyzed (Participants) | 433 | 437 | 431 | 444
  Week 26 | 0.97 (13.6) | 0.99 (14.8) | 0.98 (14.9) | 0.99 (12.6)
  Week 52: number analyzed (Participants) | 421 | 427 | 431 | 435
  Week 52 | 0.99 (13.9) | 1.01 (14.3) | 1.01 (15.2) | 0.99 (15.9)
  Week 78: number analyzed (Participants) | 419 | 419 | 420 | 438
  Week 78 | 0.97 (15.3) | 0.99 (15.6) | 1.00 (15.5) | 0.99 (14.2)

13. Secondary Outcome: Change in Triglycerides (Ratio to Baseline)
Description: Change from baseline (week 0) in triglycerides (mmol/L) at weeks 26, 52 and 78 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Ratio of triglycerides
  Week 26: number analyzed (Participants) | 433 | 437 | 431 | 444
  Week 26 | 0.99 (38.1) | 0.96 (39.2) | 0.92 (39.8) | 0.97 (36.2)
  Week 52: number analyzed (Participants) | 421 | 427 | 431 | 435
  Week 52 | 1.00 (35.7) | 0.97 (41.3) | 0.93 (42.3) | 0.98 (37.8)
  Week 78: number analyzed (Participants) | 419 | 419 | 420 | 438
  Week 78 | 0.95 (43.9) | 0.94 (43.7) | 0.92 (43.1) | 0.93 (41.6)

14. Secondary Outcome: Change in Free Fatty Acids (Ratio to Baseline)
Description: Change from baseline (week 0) in free fatty acids (FFA) (mmol/L) at weeks 26, 52 and 78 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. Because of an issue with the handling of the blood samples for FFA, all FFA data were considered invalid for this trial; thus, no conclusion with regards to FFA levels can be made based on the data presented here.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of FFA
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Ratio of FFA
  Week 26: number analyzed (Participants) | 426 | 428 | 426 | 441
  Week 26 | 0.96 (48.7) | 0.91 (50.4) | 0.88 (55.8) | 0.90 (49.8)
  Week 52: number analyzed (Participants) | 419 | 420 | 426 | 432
  Week 52 | 1.03 (46.7) | 1.00 (47.9) | 0.96 (56.0) | 0.98 (47.5)
  Week 78: number analyzed (Participants) | 415 | 413 | 414 | 435
  Week 78 | 0.92 (54.2) | 0.87 (56.5) | 0.88 (56.3) | 0.87 (57.8)

15. Secondary Outcome: Change in SMPG - Mean 7-point Profile
Description: Change from baseline (week 0) in mean 7-point self-measured plasma glucose (SMPG) profile. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. Mean 7-point profile was defined as the area under the profile, calculated using the trapezoidal method, divided by the measurement time. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
mmol/L
  Week 26: number analyzed (Participants) | 398 | 410 | 400 | 409
  Week 26 | -1.1 (2.3) | -1.5 (2.3) | -1.7 (2.4) | -1.2 (2.3)
  Week 52: number analyzed (Participants) | 399 | 405 | 401 | 414
  Week 52 | -1.3 (2.4) | -1.5 (2.5) | -1.8 (2.4) | -1.4 (2.4)
  Week 78: number analyzed (Participants) | 396 | 385 | 392 | 409
  Week 78 | -1.3 (2.7) | -1.5 (2.7) | -1.7 (2.2) | -1.3 (2.5)

16. Secondary Outcome: Change in SMPG - Mean Postprandial Increment Over All Meals
Description: Change from baseline (week 0) in the average of the post-prandial increments over all meals was evaluated at weeks 26, 52 and 78. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
mmol/L
  Week 26: number analyzed (Participants) | 400 | 411 | 402 | 408
  Week 26 | -0.4 (2.1) | -0.4 (2.1) | -0.6 (2.1) | -0.6 (2.1)
  Week 52: number analyzed (Participants) | 400 | 406 | 402 | 413
  Week 52 | -0.4 (2.0) | -0.4 (2.1) | -0.7 (2.0) | -0.4 (2.1)
  Week 78: number analyzed (Participants) | 398 | 387 | 392 | 409
  Week 78 | -0.4 (2.1) | -0.4 (2.1) | -0.6 (2.0) | -0.6 (2.2)

17. Secondary Outcome: Participants Who Achieve HbA1c <7.0% (53 mmol/Mol) ADA Target (Yes/no)
Description: Participants who achieved HbA1c <7.0% (American Diabetes Association (ADA) target) (yes/no), was evaluated at weeks 26, 52 and 78. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52, week 78
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Participants
  Week 26: number analyzed (Participants) | 435 | 438 | 436 | 446
  Week 26: Yes | 116 | 192 | 246 | 144
  Week 26: No | 319 | 246 | 190 | 302
  Week 52: number analyzed (Participants) | 427 | 431 | 434 | 436
  Week 52: Yes | 113 | 168 | 238 | 138
  Week 52: No | 314 | 263 | 196 | 298
  Week 78: number analyzed (Participants) | 421 | 424 | 425 | 439
  Week 78: Yes | 113 | 165 | 191 | 129
  Week 78: No | 308 | 259 | 234 | 310

18. Secondary Outcome: Participants Who Achieve HbA1c ≤6.5% (48 mmol/Mol) AACE Target (Yes/no)
Description: Participants who achieved HbA1c less than or equal to 6.5% (American Association of Clinical Endocrinologists (AACE) target) (yes/no) at weeks 26, 52 and 78 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52, week 78
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Participants
  Week 26: number analyzed (Participants) | 435 | 438 | 436 | 446
  Week 26: Yes | 55 | 116 | 161 | 61
  Week 26: No | 380 | 322 | 275 | 385
  Week 52: number analyzed (Participants) | 427 | 431 | 434 | 436
  Week 52: Yes | 55 | 99 | 146 | 59
  Week 52: No | 372 | 332 | 288 | 377
  Week 78: number analyzed (Participants) | 421 | 424 | 425 | 439
  Week 78: Yes | 49 | 100 | 129 | 60
  Week 78: No | 372 | 324 | 296 | 379

19. Secondary Outcome: Participants Who Achieve Weight Loss ≥5% (Yes/no)
Description: Participants who achieved weight loss more than or equal to 5% of their baseline body weight (yes/no) at weeks 26, 52 and 78 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52, week 78
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Participants
  Week 26: number analyzed (Participants) | 438 | 440 | 439 | 447
  Week 26: Yes | 53 | 81 | 131 | 45
  Week 26: No | 385 | 359 | 308 | 402
  Week 52: number analyzed (Participants) | 428 | 433 | 435 | 437
  Week 52: Yes | 66 | 118 | 147 | 50
  Week 52: No | 362 | 315 | 288 | 387
  Week 78: number analyzed (Participants) | 425 | 425 | 428 | 443
  Week 78: Yes | 83 | 115 | 139 | 59
  Week 78: No | 342 | 310 | 289 | 384

20. Secondary Outcome: Participants Who Achieve Weight Loss ≥10% (Yes/no)
Description: Participants who achieved weight loss more than or equal to 10% of their baseline body weight (yes/no) at weeks 26, 52 and 78 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52, week 78
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Participants
  Week 26: number analyzed (Participants) | 438 | 440 | 439 | 447
  Week 26: Yes | 5 | 23 | 29 | 8
  Week 26: No | 433 | 417 | 410 | 439
  Week 52: number analyzed (Participants) | 428 | 433 | 435 | 437
  Week 52: Yes | 13 | 31 | 48 | 11
  Week 52: No | 415 | 402 | 387 | 426
  Week 78: number analyzed (Participants) | 425 | 425 | 428 | 443
  Week 78: Yes | 12 | 43 | 46 | 17
  Week 78: No | 413 | 382 | 382 | 426

21. Secondary Outcome: Participants Who Achieve HbA1c <7.0 % (53 mmol/Mol) Without Hypoglycaemia (Severe or BG Confirmed Symptomatic Hypoglycaemia) and no Weight Gain (Yes/no)
Description: Participants who achieved HbA1c less than 7.0 % without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia and without weight gain (yes/no) at weeks 26, 52 and 78 are presented. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia was defined as an episode with plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52, week 78
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Participants
  Week 26: number analyzed (Participants) | 435 | 438 | 436 | 446
  Week 26: Yes | 87 | 155 | 208 | 90
  Week 26: No | 348 | 283 | 228 | 356
  Week 52: number analyzed (Participants) | 427 | 431 | 434 | 436
  Week 52: Yes | 87 | 134 | 195 | 87
  Week 52: No | 340 | 297 | 239 | 349
  Week 78: number analyzed (Participants) | 421 | 424 | 425 | 439
  Week 78: Yes | 85 | 136 | 151 | 84
  Week 78: No | 336 | 288 | 274 | 355

22. Secondary Outcome: Participants Who Achieve HbA1c Reduction ≥1% (10.9 mmol/Mol) and Weight Loss ≥3% (Yes/no)
Description: Participants who achieved HbA1c reduction more than or equal to 1% of their baseline HbA1c and weight loss of more than or equal to 3% of their baseline body weight (yes/no) at weeks 26, 52 and 78 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52, week 78
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Participants
  Week 26: number analyzed (Participants) | 435 | 438 | 436 | 446
  Week 26: Yes | 55 | 117 | 166 | 43
  Week 26: No | 380 | 321 | 270 | 403
  Week 52: number analyzed (Participants) | 427 | 431 | 434 | 436
  Week 52: Yes | 73 | 106 | 164 | 51
  Week 52: No | 354 | 325 | 270 | 385
  Week 78: number analyzed (Participants) | 421 | 424 | 425 | 439
  Week 78: Yes | 76 | 113 | 149 | 60
  Week 78: No | 345 | 311 | 276 | 379

23. Secondary Outcome: Time to Additional Anti-diabetic Medication
Description: Presented results are the number of participants who had taken additional anti-diabetic medication anytime during the periods, from week 0 to week 26, week 0 to week 52 and week 0 to week 78. Additional anti-diabetic medication was defined as any new anti-diabetic medication used for more than 21 days with the initiation at or after randomisation (week 0) and before (planned) end-of-treatment (week 78), and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before (planned) end-of-treatment. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-78
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Participants
  Week 0 to week 26 | 33 | 20 | 15 | 20
  Week 0 to week 52 | 137 | 86 | 51 | 111
  Week 0 to week 78 | 179 | 119 | 75 | 148
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Sitagliptin 100 mg; Time to initiation of additional anti-diabetic medication was analysed using a Cox proportional hazards model with treatment, strata, and region as categorical fixed effects and baseline HbA1c as covariate. Withdrawal for any reason or lost to follow-up contributed to the analysis as events (initiation of additional anti-diabetic medication). Censoring time was one day before planned end of treatment; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0063, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [1.09 to 1.65] — Oral semaglutide 3 mg / Sitagliptin 100 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Sitagliptin 100 mg; [analysis description as in outcome 23, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0221, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.61 to 0.96] — Oral semaglutide 7 mg / Sitagliptin 100 mg
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Sitagliptin 100 mg; [analysis description as in outcome 23, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.41 to 0.68] — Oral semaglutide 14 mg / Sitagliptin 100 mg

24. Secondary Outcome: Time to Rescue Medication
Description: Presented results are the number of participants who had taken rescue medication anytime during the periods, from week 0 to week 26, week 0 to week 52 and week 0 to week 78. Rescue medication was defined as any new anti-diabetic medication used as add-on to trial product and used for more than 21 days with the initiation at or after randomisation (week 0) and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before last day on trial product. Results are based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Weeks 0-78
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Participants
  Week 0 to week 26 | 25 | 11 | 5 | 13
  Week 0 to week 52 | 121 | 73 | 31 | 94
  Week 0 to week 78 | 160 | 103 | 47 | 129
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Sitagliptin 100 mg; Time to initiation of rescue medication was analysed using a Cox proportional hazards model with treatment, strata, and region as categorical fixed effects and baseline HbA1c as covariate. Censoring time was one day before last day on trial product; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0160, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [1.05 to 1.68] — Oral semaglutide 3 mg / Sitagliptin 100 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Sitagliptin 100 mg; [analysis description as in outcome 24, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0022, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.51 to 0.86] — Oral semaglutide 7 mg / Sitagliptin 100 mg
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Sitagliptin 100 mg; [analysis description as in outcome 24, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.22 to 0.43] — Oral semaglutide 14 mg / Sitagliptin 100 mg

25. Secondary Outcome: Number of TEAEs During Exposure to Trial Product
Description: Treatment emergent adverse events (TEAEs) were recorded from week 0 to week 83 (78-week treatment period plus the 5-week follow-up period). Adverse events (AEs) with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period: Time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-83
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 464 | 465 | 466
Events | 1774 | 1686 | 1824 | 1852

26. Secondary Outcome: Change in Amylase (Ratio to Baseline)
Description: Change from baseline (week 0) in amylase (units/litre (U/L)) at weeks 26, 52 and 78 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52, week 78
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product. Number Analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 464 | 465 | 466
Ratio
  Week 26: number analyzed (Participants) | 415 | 421 | 401 | 433
  Week 26 | 1.03 (25.6) | 1.07 (27.5) | 1.14 (30.4) | 1.08 (21.4)
  Week 52: number analyzed (Participants) | 391 | 403 | 388 | 414
  Week 52 | 1.03 (25.8) | 1.09 (28.8) | 1.11 (29.0) | 1.08 (24.1)
  Week 78: number analyzed (Participants) | 377 | 392 | 366 | 402
  Week 78 | 1.02 (28.4) | 1.09 (29.2) | 1.09 (25.5) | 1.08 (25.9)

27. Secondary Outcome: Change in Lipase (Ratio to Baseline)
Description: Change from baseline (week 0) in lipase (U/L) at weeks 26, 52 and 78 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 464 | 465 | 466
Ratio
  Week 26: number analyzed (Participants) | 415 | 420 | 401 | 433
  Week 26 | 1.07 (52.6) | 1.13 (60.1) | 1.26 (64.9) | 1.14 (50.3)
  Week 52: number analyzed (Participants) | 391 | 403 | 388 | 414
  Week 52 | 1.06 (51.5) | 1.15 (59.4) | 1.25 (56.6) | 1.15 (54.2)
  Week 78: number analyzed (Participants) | 377 | 392 | 366 | 402
  Week 78 | 1.04 (56.2) | 1.14 (61.9) | 1.18 (54.3) | 1.10 (50.7)

28. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline (week 0) in pulse rate was evaluated at weeks 26, 52 and 78. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 464 | 465 | 466
Beats/minute
  Week 26: number analyzed (Participants) | 419 | 422 | 406 | 435
  Week 26 | 1 (9) | 2 (9) | 3 (10) | 0 (10)
  Week 52: number analyzed (Participants) | 396 | 406 | 391 | 416
  Week 52 | 0 (10) | 2 (9) | 2 (10) | -0 (10)
  Week 78: number analyzed (Participants) | 382 | 394 | 368 | 405
  Week 78 | 1 (10) | 1 (10) | 2 (10) | 0 (10)

29. Secondary Outcome: Change in SBP and DBP
Description: Change from baseline (week 0) in systolic blood pressure (SBP) and diastolic blood pressure (DBP) was evaluated at weeks 26, 52 and 78. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 464 | 465 | 466
mmHg
  SBP: Week 26: number analyzed (Participants) | 419 | 422 | 406 | 435
  SBP: Week 26 | -2 (14) | -2 (15) | -3 (14) | -2 (15)
  SBP: Week 52: number analyzed (Participants) | 397 | 406 | 391 | 416
  SBP: Week 52 | -2 (15) | -4 (14) | -3 (15) | -1 (14)
  SBP: Week 78: number analyzed (Participants) | 382 | 394 | 369 | 405
  SBP: Week 78 | -2 (15) | -3 (15) | -3 (14) | 0 (15)
  DBP: Week 26: number analyzed (Participants) | 419 | 422 | 406 | 435
  DBP: Week 26 | -1 (9) | -0 (9) | -1 (9) | -0 (9)
  DBP: Week 52: number analyzed (Participants) | 397 | 406 | 391 | 416
  DBP: Week 52 | -2 (9) | -1 (9) | -1 (9) | -1 (9)
  DBP: Week 78: number analyzed (Participants) | 382 | 394 | 369 | 405
  DBP: Week 78 | -1 (10) | -1 (10) | -1 (10) | -1 (10)

30. Secondary Outcome: Change in ECG Evaluation
Description: Change from baseline (week 0) in electrocardiogram (ECG) was evaluated at weeks 26, 52 and 78. Change from baseline results are presented as shift in findings (normal, abnormal and not clinically significant (NCS) and abnormal and clinically significant (CS)) from week 0 to week 26, 52 and 78. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 464 | 465 | 466
Participants
  Normal (week 0) to normal (week 26): number analyzed (Participants) | 253 | 261 | 254 | 249
  Normal (week 0) to normal (week 26) | 211 | 214 | 230 | 204
  Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 253 | 261 | 254 | 249
  Normal (week 0) to abnormal NCS (week 26) | 38 | 42 | 24 | 41
  Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 253 | 261 | 254 | 249
  Normal (week 0) to abnormal CS (week 26) | 4 | 5 | 0 | 4
  Abnormal (week 0) NCS to normal (week 26): number analyzed (Participants) | 177 | 173 | 176 | 186
  Abnormal (week 0) NCS to normal (week 26) | 41 | 44 | 42 | 40
  Abnormal (week 0) NCS to abnormal NCS (week 26): number analyzed (Participants) | 177 | 173 | 176 | 186
  Abnormal (week 0) NCS to abnormal NCS (week 26) | 132 | 128 | 133 | 143
  Abnormal (week 0) NCS to abnormal CS (week 26): number analyzed (Participants) | 177 | 173 | 176 | 186
  Abnormal (week 0) NCS to abnormal CS (week 26) | 4 | 1 | 1 | 3
  Abnormal (week 0) CS to normal (week 26): number analyzed (Participants) | 8 | 5 | 9 | 9
  Abnormal (week 0) CS to normal (week 26) | 1 | 1 | 0 | 3
  Abnormal (week 0) CS to abnormal NCS (week 26): number analyzed (Participants) | 8 | 5 | 9 | 9
  Abnormal (week 0) CS to abnormal NCS (week 26) | 3 | 2 | 3 | 2
  Abnormal (week 0) CS to abnormal CS (week 26): number analyzed (Participants) | 8 | 5 | 9 | 9
  Abnormal (week 0) CS to abnormal CS (week 26) | 4 | 2 | 6 | 4
  Normal (week 0) to normal (week 52): number analyzed (Participants) | 244 | 255 | 253 | 248
  Normal (week 0) to normal (week 52) | 196 | 218 | 219 | 204
  Normal (week 0) to abnormal NCS (week 52): number analyzed (Participants) | 244 | 255 | 253 | 248
  Normal (week 0) to abnormal NCS (week 52) | 47 | 37 | 33 | 40
  Normal (week 0) to abnormal CS (week 52): number analyzed (Participants) | 244 | 255 | 253 | 248
  Normal (week 0) to abnormal CS (week 52) | 1 | 0 | 1 | 4
  Abnormal (week 0) NCS to normal (week 52): number analyzed (Participants) | 175 | 173 | 174 | 178
  Abnormal (week 0) NCS to normal (week 52) | 40 | 49 | 56 | 48
  Abnormal (week 0) NCS to abnormal NCS (week 52): number analyzed (Participants) | 175 | 173 | 174 | 178
  Abnormal (week 0) NCS to abnormal NCS (week 52) | 131 | 123 | 118 | 128
  Abnormal (week 0) NCS to abnormal CS (week 52): number analyzed (Participants) | 175 | 173 | 174 | 178
  Abnormal (week 0) NCS to abnormal CS (week 52) | 4 | 1 | 0 | 2
  Abnormal (week 0) CS to normal (week 52): number analyzed (Participants) | 8 | 5 | 9 | 9
  Abnormal (week 0) CS to normal (week 52) | 1 | 1 | 2 | 1
  Abnormal (week 0) CS to abnormal NCS (week 52): number analyzed (Participants) | 8 | 5 | 9 | 9
  Abnormal (week 0) CS to abnormal NCS (week 52) | 3 | 3 | 0 | 2
  Abnormal (week 0) CS to abnormal CS (week 52): number analyzed (Participants) | 8 | 5 | 9 | 9
  Abnormal (week 0) CS to abnormal CS (week 52) | 4 | 1 | 7 | 6
  Normal (week 0) to normal (week 78): number analyzed (Participants) | 240 | 246 | 251 | 249
  Normal (week 0) to normal (week 78) | 196 | 201 | 219 | 208
  Normal (week 0) to abnormal NCS (week 78): number analyzed (Participants) | 240 | 246 | 251 | 249
  Normal (week 0) to abnormal NCS (week 78) | 41 | 43 | 31 | 40
  Normal (week 0) to abnormal CS (week 78): number analyzed (Participants) | 240 | 246 | 251 | 249
  Normal (week 0) to abnormal CS (week 78) | 3 | 2 | 1 | 1
  Abnormal (week 0) NCS to normal (week 78): number analyzed (Participants) | 175 | 171 | 168 | 182
  Abnormal (week 0) NCS to normal (week 78) | 39 | 45 | 51 | 47
  Abnormal (week 0) NCS to abnormal NCS (week 78): number analyzed (Participants) | 175 | 171 | 168 | 182
  Abnormal (week 0) NCS to abnormal NCS (week 78) | 131 | 125 | 114 | 133
  Abnormal (week 0) NCS to abnormal CS (week 78): number analyzed (Participants) | 175 | 171 | 168 | 182
  Abnormal (week 0) NCS to abnormal CS (week 78) | 5 | 1 | 3 | 2
  Abnormal (week 0) CS to normal (week 78): number analyzed (Participants) | 8 | 6 | 9 | 9
  Abnormal (week 0) CS to normal (week 78) | 0 | 3 | 1 | 3
  Abnormal (week 0) CS to abnormal NCS (week 78): number analyzed (Participants) | 8 | 6 | 9 | 9
  Abnormal (week 0) CS to abnormal NCS (week 78) | 4 | 2 | 3 | 2
  Abnormal (week 0) CS to abnormal CS (week 78): number analyzed (Participants) | 8 | 6 | 9 | 9
  Abnormal (week 0) CS to abnormal CS (week 78) | 4 | 1 | 5 | 4

31. Secondary Outcome: Change in Physical Examination
Description: Participants with physical examination findings, normal, abnormal NCS and abnormal CS at baseline (weeks -2), weeks 52 and 78 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. Results are presented for the following examinations: 1) Cardiovascular system; 2) Central and peripheral nervous system; 3) Gastrointestinal system, incl. mouth; 4) General appearance; 5) Head, ears, eyes, nose, throat, neck; 6) Lymph node palpation; 7) Musculoskeletal system; 8) Respiratory system; 9) Skin; 10) Thyroid gland.
Time Frame: Week -2, week 52, week 78
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 464 | 465 | 466
Participants
  1) Cardiovascular system (week -2): Normal | 431 | 425 | 432 | 424
  1) Cardiovascular system (week -2): Abnormal NCS | 30 | 38 | 30 | 41
  1) Cardiovascular system (week -2): Abnormal CS | 5 | 1 | 3 | 1
  1) Cardiovascular system (week 52): number analyzed (Participants) | 427 | 433 | 435 | 436
  1) Cardiovascular system (week 52): Normal | 398 | 396 | 404 | 399
  1) Cardiovascular system (week 52): Abnormal NCS | 24 | 36 | 28 | 37
  1) Cardiovascular system (week 52): Abnormal CS | 5 | 1 | 3 | 0
  1) Cardiovascular system (week 78): number analyzed (Participants) | 424 | 423 | 428 | 441
  1) Cardiovascular system (week 78): Normal | 395 | 386 | 402 | 399
  1) Cardiovascular system (week 78): Abnormal NCS | 24 | 33 | 24 | 41
  1) Cardiovascular system (week 78): Abnormal CS | 5 | 4 | 2 | 1
  2) Central and peripheral nervous system (week -2): number analyzed (Participants) | 466 | 463 | 464 | 466
  2) Central and peripheral nervous system (week -2): Normal | 410 | 415 | 407 | 409
  2) Central and peripheral nervous system (week -2): Abnormal NCS | 44 | 42 | 49 | 43
  2) Central and peripheral nervous system (week -2): Abnormal CS | 12 | 6 | 8 | 14
  2) Central and peripheral nervous system (week 52): number analyzed (Participants) | 427 | 433 | 435 | 435
  2) Central and peripheral nervous system (week 52): Normal | 376 | 382 | 388 | 385
  2) Central and peripheral nervous system (week 52): Abnormal NCS | 44 | 45 | 38 | 42
  2) Central and peripheral nervous system (week 52): Abnormal CS | 7 | 6 | 9 | 8
  2) Central and peripheral nervous system (week 78): number analyzed (Participants) | 424 | 423 | 428 | 441
  2) Central and peripheral nervous system (week 78): Normal | 377 | 376 | 384 | 399
  2) Central and peripheral nervous system (week 78): Abnormal NCS | 43 | 43 | 37 | 37
  2) Central and peripheral nervous system (week 78): Abnormal CS | 4 | 4 | 7 | 5
  3) Gastrointestinal system, incl. mouth (week -2): Normal | 419 | 421 | 420 | 421
  3) Gastrointestinal system, incl. mouth (week -2): Abnormal NCS | 45 | 39 | 45 | 45
  3) Gastrointestinal system, incl. mouth (week -2): Abnormal CS | 2 | 4 | 0 | 0
  3) Gastrointestinal system, incl. mouth (week 52): number analyzed (Participants) | 426 | 433 | 435 | 436
  3) Gastrointestinal system, incl. mouth (week 52): Normal | 386 | 402 | 397 | 394
  3) Gastrointestinal system, incl. mouth (week 52): Abnormal NCS | 39 | 28 | 36 | 40
  3) Gastrointestinal system, incl. mouth (week 52): Abnormal CS | 1 | 3 | 2 | 2
  3) Gastrointestinal system, incl. mouth (week 78): number analyzed (Participants) | 424 | 423 | 428 | 441
  3) Gastrointestinal system, incl. mouth (week 78): Normal | 398 | 387 | 393 | 408
  3) Gastrointestinal system, incl. mouth (week 78): Abnormal NCS | 26 | 31 | 35 | 31
  3) Gastrointestinal system, incl. mouth (week 78): Abnormal CS | 0 | 5 | 0 | 2
  4) General appearance (week -2): Normal | 407 | 405 | 412 | 405
  4) General appearance (week -2): Abnormal NCS | 43 | 45 | 38 | 46
  4) General appearance (week -2): Abnormal CS | 16 | 14 | 15 | 15
  4) General appearance (week 52): number analyzed (Participants) | 426 | 433 | 435 | 436
  4) General appearance (week 52): Normal | 381 | 384 | 390 | 385
  4) General appearance (week 52): Abnormal NCS | 37 | 37 | 33 | 39
  4) General appearance (week 52): Abnormal CS | 8 | 12 | 12 | 12
  4) General appearance (week 78): number analyzed (Participants) | 424 | 423 | 428 | 441
  4) General appearance (week 78): Normal | 379 | 373 | 388 | 394
  4) General appearance (week 78): Abnormal NCS | 37 | 40 | 28 | 37
  4) General appearance (week 78): Abnormal CS | 8 | 10 | 12 | 10
  5) Head, ears, eyes, nose, throat, neck (week -2): Normal | 441 | 440 | 435 | 444
  5) Head, ears, eyes, nose, throat, neck (week -2): Abnormal NCS | 25 | 24 | 27 | 21
  5) Head, ears, eyes, nose, throat, neck (week -2): Abnormal CS | 0 | 0 | 3 | 1
  5) Head, ears, eyes, nose, throat, neck (week 52): number analyzed (Participants) | 426 | 433 | 435 | 436
  5) Head, ears, eyes, nose, throat, neck (week 52): Normal | 398 | 411 | 404 | 410
  5) Head, ears, eyes, nose, throat, neck (week 52): Abnormal NCS | 25 | 21 | 27 | 26
  5) Head, ears, eyes, nose, throat, neck (week 52): Abnormal CS | 3 | 1 | 4 | 0
  5) Head, ears, eyes, nose, throat, neck (week 78): number analyzed (Participants) | 424 | 423 | 428 | 441
  5) Head, ears, eyes, nose, throat, neck (week 78): Normal | 400 | 405 | 399 | 415
  5) Head, ears, eyes, nose, throat, neck (week 78): Abnormal NCS | 22 | 17 | 28 | 25
  5) Head, ears, eyes, nose, throat, neck (week 78): Abnormal CS | 2 | 1 | 1 | 1
  6) Lymph node palpation (week -2): number analyzed (Participants) | 466 | 463 | 465 | 466
  6) Lymph node palpation (week -2): Normal | 466 | 462 | 463 | 464
  6) Lymph node palpation (week -2): Abnormal NCS | 0 | 1 | 2 | 2
  6) Lymph node palpation (week -2): Abnormal CS | 0 | 0 | 0 | 0
  6) Lymph node palpation (week 52): number analyzed (Participants) | 426 | 433 | 435 | 436
  6) Lymph node palpation (week 52): Normal | 425 | 432 | 434 | 436
  6) Lymph node palpation (week 52): Abnormal NCS | 1 | 1 | 1 | 0
  6) Lymph node palpation (week 52): Abnormal CS | 0 | 0 | 0 | 0
  6) Lymph node palpation (week 78): number analyzed (Participants) | 423 | 423 | 428 | 441
  6) Lymph node palpation (week 78): Normal | 421 | 423 | 425 | 441
  6) Lymph node palpation (week 78): Abnormal NCS | 2 | 0 | 3 | 0
  6) Lymph node palpation (week 78): Abnormal CS | 0 | 0 | 0 | 0
  7) Musculoskeletal system (week -2): Normal | 421 | 435 | 440 | 430
  7) Musculoskeletal system (week -2): Abnormal NCS | 39 | 24 | 23 | 32
  7) Musculoskeletal system (week -2): Abnormal CS | 6 | 5 | 2 | 4
  7) Musculoskeletal system (week 52): number analyzed (Participants) | 426 | 433 | 435 | 435
  7) Musculoskeletal system (week 52): Normal | 383 | 400 | 408 | 403
  7) Musculoskeletal system (week 52): Abnormal NCS | 37 | 28 | 24 | 26
  7) Musculoskeletal system (week 52): Abnormal CS | 6 | 5 | 3 | 6
  7) Musculoskeletal system (week 78): number analyzed (Participants) | 424 | 423 | 428 | 441
  7) Musculoskeletal system (week 78): Normal | 388 | 389 | 402 | 413
  7) Musculoskeletal system (week 78): Abnormal NCS | 33 | 31 | 24 | 23
  7) Musculoskeletal system (week 78): Abnormal CS | 3 | 3 | 2 | 5
  8) Respiratory system (week -2): Normal | 458 | 451 | 462 | 456
  8) Respiratory system (week -2): Abnormal NCS | 6 | 9 | 2 | 10
  8) Respiratory system (week -2): Abnormal CS | 2 | 4 | 1 | 0
  8) Respiratory system (week 52): number analyzed (Participants) | 426 | 433 | 435 | 436
  8) Respiratory system (week 52): Normal | 418 | 427 | 431 | 429
  8) Respiratory system (week 52): Abnormal NCS | 6 | 4 | 3 | 6
  8) Respiratory system (week 52): Abnormal CS | 2 | 2 | 1 | 1
  8) Respiratory system (week 78): number analyzed (Participants) | 424 | 423 | 428 | 441
  8) Respiratory system (week 78): Normal | 419 | 418 | 427 | 434
  8) Respiratory system (week 78): Abnormal NCS | 3 | 4 | 1 | 6
  8) Respiratory system (week 78): Abnormal CS | 2 | 1 | 0 | 1
  9) Skin (week -2): Normal | 394 | 400 | 394 | 402
  9) Skin (week -2): Abnormal NCS | 66 | 56 | 61 | 58
  9) Skin (week -2): Abnormal CS | 6 | 8 | 10 | 6
  9) Skin (week 52): number analyzed (Participants) | 427 | 433 | 435 | 436
  9) Skin (week 52): Normal | 372 | 383 | 383 | 375
  9) Skin (week 52): Abnormal NCS | 52 | 44 | 44 | 51
  9) Skin (week 52): Abnormal CS | 3 | 6 | 8 | 10
  9) Skin (week 78): number analyzed (Participants) | 424 | 423 | 428 | 441
  9) Skin (week 78): Normal | 361 | 370 | 382 | 393
  9) Skin (week 78): Abnormal NCS | 55 | 45 | 38 | 41
  9) Skin (week 78): Abnormal CS | 8 | 8 | 8 | 7
  10) Thyroid gland (week -2): number analyzed (Participants) | 465 | 464 | 465 | 466
  10) Thyroid gland (week -2): Normal | 451 | 452 | 451 | 454
  10) Thyroid gland (week -2): Abnormal NCS | 13 | 11 | 11 | 12
  10) Thyroid gland (week -2): Abnormal CS | 1 | 1 | 3 | 0
  10) Thyroid gland (week 52): number analyzed (Participants) | 426 | 433 | 435 | 436
  10) Thyroid gland (week 52): Normal | 413 | 423 | 425 | 427
  10) Thyroid gland (week 52): Abnormal NCS | 11 | 10 | 7 | 8
  10) Thyroid gland (week 52): Abnormal CS | 2 | 0 | 3 | 1
  10) Thyroid gland (week 78): number analyzed (Participants) | 424 | 423 | 428 | 441
  10) Thyroid gland (week 78): Normal | 411 | 411 | 418 | 433
  10) Thyroid gland (week 78): Abnormal NCS | 11 | 12 | 8 | 7
  10) Thyroid gland (week 78): Abnormal CS | 2 | 0 | 2 | 1

32. Secondary Outcome: Change in Eye Examination Category
Description: Participants with eye examination (fundoscopy) findings, normal, abnormal NCS and abnormal CS at baseline (week -2), week 52 and week 78 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week -2, week 52, week 78
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 464 | 465 | 466
Participants
  Left eye (week -2): number analyzed (Participants) | 459 | 455 | 457 | 463
  Left eye (week -2): Normal | 302 | 299 | 305 | 297
  Left eye (week -2): Abnormal NCS | 130 | 138 | 129 | 137
  Left eye (week -2): Abnormal CS | 27 | 18 | 23 | 29
  Left eye (week 52): number analyzed (Participants) | 393 | 388 | 391 | 405
  Left eye (week 52): Normal | 249 | 253 | 270 | 252
  Left eye (week 52): Abnormal NCS | 119 | 113 | 101 | 126
  Left eye (week 52): Abnormal CS | 25 | 22 | 20 | 27
  Left eye (week 78): number analyzed (Participants) | 417 | 415 | 420 | 431
  Left eye (week 78): Normal | 261 | 255 | 273 | 287
  Left eye (week 78): Abnormal NCS | 135 | 141 | 130 | 113
  Left eye (week 78): Abnormal CS | 21 | 19 | 17 | 31
  Right eye (week -2): number analyzed (Participants) | 459 | 454 | 457 | 463
  Right eye (week -2): Normal | 309 | 298 | 308 | 297
  Right eye (week -2): Abnormal NCS | 126 | 139 | 126 | 138
  Right eye (week -2): Abnormal CS | 24 | 17 | 23 | 28
  Right eye (week 52): number analyzed (Participants) | 393 | 388 | 391 | 405
  Right eye (week 52): Normal | 247 | 256 | 271 | 255
  Right eye (week 52): Abnormal NCS | 122 | 112 | 103 | 123
  Right eye (week 52): Abnormal CS | 24 | 20 | 17 | 27
  Right eye (week 78): number analyzed (Participants) | 417 | 415 | 420 | 431
  Right eye (week 78): Normal | 258 | 255 | 275 | 279
  Right eye (week 78): Abnormal NCS | 136 | 146 | 128 | 122
  Right eye (week 78): Abnormal CS | 23 | 14 | 17 | 30

33. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). Number of participants who measured with anti-semaglutide binding antibodies anytime during post-baseline visits (weeks 0-83) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-83
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 459 | 460 | 465
Participants | 1 | 2 | 3

34. Secondary Outcome: Occurrence of Anti-semaglutide Neutralising Antibodies (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). Number of participants who measured with anti-semaglutide neutralising antibodies anytime during post-baseline visits (weeks 0-83) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-83
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 459 | 460 | 465
Participants | 0 | 0 | 0

35. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). Number of participants who measured with anti-semaglutide binding antibodies cross reacting with native glucagon-like peptide-1 (GLP-1) anytime during post-baseline visits (weeks 0-83) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-83
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 459 | 460 | 465
Participants | 0 | 1 | 1

36. Secondary Outcome: Occurrence of Anti-semaglutide Neutralising Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). Number of participants who measured with anti-semaglutide neutralising antibodies cross reacting with native GLP-1 anytime during post-baseline visits (weeks 0-83) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-83
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 459 | 460 | 465
Participants | 0 | 0 | 0

37. Secondary Outcome: Anti-semaglutide Binding Antibody Levels
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). It is based on the data from participants who were measured with anti-semaglutide antibodies anytime during post-baseline visits (weeks 0-83). Results are presented as percentage of bound radioactivity-labelled semaglutide /total added radioactivity-labelled semaglutide (%B/T). Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-83
Population: Overall number of participants analysed = participants who were found positive for anti-semaglutide antibodies.
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 1 | 2 | 3
%B/T
  Week 4: number analyzed (Participants) | 0 | 0 | 1
  Week 4 |  |  | 9.82 (0)
  Week 8: number analyzed (Participants) | 1 | 0 | 0
  Week 8 | 1.93 (0) |  |
  Week 14: number analyzed (Participants) | 0 | 1 | 0
  Week 14 |  | 3.28 (0) |
  Week 26: number analyzed (Participants) | 0 | 1 | 1
  Week 26 |  | 2.39 (0) | 2.05 (0)
  Week 38: number analyzed (Participants) | 0 | 0 | 1
  Week 38 |  |  | 2.24 (0)
  Week 52: number analyzed (Participants) | 0 | 0 | 0
  Week 78: number analyzed (Participants) | 0 | 0 | 0
  Week 83: number analyzed (Participants) | 0 | 0 | 0

38. Secondary Outcome: Number of Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded during weeks 0-83 (78-week treatment period plus the 5-week follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a subject was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-83
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 464 | 465 | 466
Episodes | 56 | 42 | 60 | 76

39. Secondary Outcome: Participants With Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded from week 0 to week 83 (78-week treatment period plus the 5-week follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a subject was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-83
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 464 | 465 | 466
Participants | 23 | 24 | 36 | 39

40. Secondary Outcome: Semaglutide Plasma Concentration in a Subset of the Participants for Population PK Analyses
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). Semaglutide plasma concentrations for participants in the pharmacokinetic (PK) subpopulation are presented. The PK subpopulation consisted of participants from sites in Germany, Japan and the United States receiving oral semaglutide (3 mg, 7 mg or 14 mg). Results are based on the data from the on-treatment observation period and follow-up period. The on-treatment observation period was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-83
Population: Overall number of participants analysed = number of participants in the PK subpopulation. Number Analyzed = number of participants with available data in the PK subpopulation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 221 | 215 | 205
nmol/L
  Week 0: number analyzed (Participants) | 193 | 187 | 179
  Week 0 | 0.4 (0.0) | 0.4 (0.0) | 0.4 (0.0)
  Week 4: number analyzed (Participants) | 212 | 208 | 197
  Week 4 | 1.5 (109.3) | 1.5 (102.1) | 1.6 (109.1)
  Week 8: number analyzed (Participants) | 208 | 198 | 190
  Week 8 | 1.5 (103.9) | 4.1 (129.4) | 4.2 (128.0)
  Week 14: number analyzed (Participants) | 201 | 190 | 185
  Week 14 | 1.4 (111.8) | 4.0 (146.8) | 9.4 (156.6)
  Week 26: number analyzed (Participants) | 191 | 190 | 171
  Week 26 | 1.3 (104.5) | 3.7 (122.5) | 8.6 (162.2)
  Week 38: number analyzed (Participants) | 183 | 180 | 168
  Week 38 | 1.4 (107.8) | 3.5 (106.4) | 8.6 (163.0)
  Week 52: number analyzed (Participants) | 176 | 178 | 165
  Week 52 | 1.4 (105.8) | 3.5 (119.0) | 8.2 (167.0)
  Week 78: number analyzed (Participants) | 167 | 173 | 155
  Week 78 | 1.3 (115.3) | 3.5 (127.2) | 8.9 (152.7)
  Week 83: number analyzed (Participants) | 165 | 172 | 154
  Week 83 | 0.4 (10.3) | 0.4 (16.5) | 0.4 (42.6)

41. Secondary Outcome: Change in SF-36v2 (Acute Version) Health Survey: Scores From the 8 Domains, the Physical Component Summary (PCS) and the Mental Component Summary (MCS)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from baseline (week 0) in the domain scores and component summary (PCS and MCS) scores were evaluated at weeks 26, 52 and 78. A positive change score indicates an improvement since baseline. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Score on a scale
  1) Physical functioning (week 26): number analyzed (Participants) | 438 | 438 | 437 | 447
  1) Physical functioning (week 26) | 0.37 (7.25) | 1.12 (6.52) | 0.63 (7.13) | 0.46 (6.73)
  1) Physical functioning (week 52): number analyzed (Participants) | 428 | 433 | 434 | 437
  1) Physical functioning (week 52) | 0.29 (7.14) | 0.64 (7.34) | 0.36 (7.30) | 0.06 (7.30)
  1) Physical functioning (week 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  1) Physical functioning (week 78) | 0.06 (8.09) | 0.94 (6.91) | 0.54 (7.98) | 0.09 (7.60)
  2) Role-Physical (week 26): number analyzed (Participants) | 438 | 438 | 437 | 447
  2) Role-Physical (week 26) | 0.42 (7.85) | 0.76 (7.15) | -0.13 (7.59) | 0.38 (8.00)
  2) Role-Physical (week 52): number analyzed (Participants) | 428 | 433 | 434 | 437
  2) Role-Physical (week 52) | -0.05 (8.40) | -0.06 (9.42) | -0.82 (8.49) | -0.69 (8.08)
  2) Role-Physical (week 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  2) Role-Physical (week 78) | 0.28 (8.14) | -0.01 (8.40) | -0.33 (7.57) | 0.44 (7.96)
  3) Bodily pain (week 26): number analyzed (Participants) | 438 | 438 | 437 | 447
  3) Bodily pain (week 26) | 0.56 (9.20) | -0.11 (8.60) | 0.22 (9.02) | 0.44 (9.18)
  3) Bodily pain (week 52): number analyzed (Participants) | 428 | 433 | 433 | 437
  3) Bodily pain (week 52) | 0.16 (9.44) | -0.65 (9.92) | -0.64 (9.40) | 0.67 (8.93)
  3) Bodily pain (week 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  3) Bodily pain (week 78) | 0.48 (9.24) | 0.32 (8.85) | 0.74 (9.40) | 0.54 (9.44)
  4) General health (week 26): number analyzed (Participants) | 438 | 438 | 437 | 447
  4) General health (week 26) | 1.17 (6.50) | 1.67 (6.98) | 1.19 (7.00) | 1.42 (7.02)
  4) General health (week 52): number analyzed (Participants) | 428 | 433 | 434 | 437
  4) General health (week 52) | 1.06 (7.07) | 1.20 (7.08) | 1.03 (6.88) | 0.95 (7.38)
  4) General health (week 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  4) General health (week 78) | 1.02 (7.23) | 1.21 (7.60) | 1.21 (7.62) | 1.32 (7.99)
  5) Vitality (week 26): number analyzed (Participants) | 438 | 438 | 437 | 447
  5) Vitality (week 26) | 0.59 (7.28) | 1.11 (7.30) | 0.88 (7.42) | 1.03 (7.42)
  5) Vitality (week 52): number analyzed (Participants) | 428 | 433 | 434 | 437
  5) Vitality (week 52) | 0.45 (7.50) | 0.79 (8.33) | 0.58 (8.15) | 0.19 (7.73)
  5) Vitality (week 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  5) Vitality (week 78) | 1.05 (8.06) | 0.85 (7.92) | 0.71 (8.42) | 1.07 (8.27)
  6) Social functioning (week 26): number analyzed (Participants) | 438 | 438 | 437 | 447
  6) Social functioning (week 26) | 0.11 (7.93) | 0.15 (8.03) | 0.31 (7.33) | 0.09 (8.38)
  6) Social functioning (week 52): number analyzed (Participants) | 428 | 433 | 434 | 437
  6) Social functioning (week 52) | -0.25 (8.35) | -0.37 (9.39) | -0.83 (8.83) | -0.68 (9.23)
  6) Social functioning (week 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  6) Social functioning (week 78) | -0.38 (8.29) | 0.19 (8.77) | -0.27 (8.66) | 0.57 (8.93)
  7) Role emotional (week 26): number analyzed (Participants) | 438 | 438 | 437 | 447
  7) Role emotional (week 26) | 0.84 (10.47) | 0.67 (9.18) | -0.37 (9.77) | 0.15 (9.97)
  7) Role emotional (week 52): number analyzed (Participants) | 428 | 433 | 434 | 437
  7) Role emotional (week 52) | 0.15 (10.99) | -0.45 (11.89) | -0.86 (10.65) | -0.63 (10.33)
  7) Role emotional (week 78): number analyzed (Participants) | 424 | 424 | 427 | 441
  7) Role emotional (week 78) | 0.32 (10.98) | 0.23 (10.95) | -0.30 (11.00) | -0.24 (10.58)
  8) Mental health (week 26): number analyzed (Participants) | 438 | 438 | 437 | 447
  8) Mental health (week 26) | 0.33 (8.32) | 0.24 (8.17) | 0.24 (8.14) | 0.61 (8.03)
  8) Mental health (week 52): number analyzed (Participants) | 428 | 433 | 434 | 437
  8) Mental health (week 52) | 0.45 (8.02) | 0.42 (9.11) | 0.05 (7.99) | 0.23 (8.20)
  8) Mental health (week 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  8) Mental health (week 78) | 0.19 (9.08) | 0.29 (9.33) | 0.28 (8.87) | 0.30 (9.33)
  Physical component summary (week 26): number analyzed (Participants) | 438 | 438 | 437 | 447
  Physical component summary (week 26) | 0.56 (6.42) | 0.98 (5.72) | 0.63 (6.00) | 0.69 (6.24)
  Physical component summary (week 52): number analyzed (Participants) | 428 | 433 | 434 | 437
  Physical component summary (week 52) | 0.31 (6.50) | 0.36 (6.82) | 0.09 (6.47) | 0.31 (6.54)
  Physical component summary (week 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  Physical component summary (week 78) | 0.46 (6.74) | 0.71 (6.24) | 0.67 (6.29) | 0.70 (6.38)
  Mental component summary (week 26): number analyzed (Participants) | 438 | 438 | 437 | 447
  Mental component summary (week 26) | 0.48 (8.62) | 0.34 (8.26) | 0.08 (8.18) | 0.41 (8.16)
  Mental component summary (week 52): number analyzed (Participants) | 428 | 433 | 434 | 437
  Mental component summary (week 52) | 0.23 (8.41) | -0.00 (9.43) | -0.37 (8.64) | -0.31 (8.71)
  Mental component summary (week 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  Mental component summary (week 78) | 0.27 (9.18) | 0.23 (9.50) | -0.07 (9.31) | 0.30 (9.46)

42. Secondary Outcome: Change in IWQoL-Lite-CT: Total Score and Scores From the 4 Domains
Description: The Impact of Weight on Quality of Life Clinical Trials Version (IWQOL-Lite-CT) is designed to assess the impact of changes in weight on patients' quality of life within the context of clinical trials. The items of the IWQOL-Lite-CT pertain to physical functioning (physical, physical function and pain/discomfort) and psychosocial domains and all items employ a 5-point graded response scale (never, rarely, sometimes, usually, always; or not at all true, a little true, moderately true, mostly true, completely true). All IWQOL-Lite-CT composite scores range from 0 to 100, with higher scores reflecting better levels of functioning. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Score on a scale
  1) Physical (week 26): number analyzed (Participants) | 438 | 437 | 437 | 447
  1) Physical (week 26) | 3.25 (14.81) | 2.38 (14.87) | 2.87 (17.32) | 1.97 (15.07)
  1) Physical (week 52): number analyzed (Participants) | 428 | 432 | 433 | 437
  1) Physical (week 52) | 1.84 (15.80) | 3.03 (16.32) | 3.18 (18.40) | 1.49 (16.11)
  1) Physical (week 78): number analyzed (Participants) | 425 | 425 | 427 | 441
  1) Physical (week 78) | 2.71 (16.16) | 3.55 (16.47) | 3.86 (17.37) | 2.86 (17.55)
  2) Physical function (week 26): number analyzed (Participants) | 438 | 437 | 437 | 447
  2) Physical function (week 26) | 3.52 (16.48) | 2.78 (16.13) | 3.20 (18.48) | 1.70 (16.54)
  2) Physical function (week 52): number analyzed (Participants) | 428 | 432 | 433 | 437
  2) Physical function (week 52) | 2.28 (17.00) | 3.24 (18.17) | 3.19 (19.76) | 1.22 (18.21)
  2) Physical function (week 78): number analyzed (Participants) | 425 | 425 | 427 | 441
  2) Physical function (week 78) | 2.55 (17.86) | 4.04 (17.99) | 3.76 (18.78) | 2.54 (18.96)
  3) Pain/discomfort (week 26): number analyzed (Participants) | 438 | 437 | 437 | 447
  3) Pain/discomfort (week 26) | 2.51 (20.28) | 1.37 (21.34) | 2.03 (22.10) | 2.66 (21.27)
  3) Pain/discomfort (week 52): number analyzed (Participants) | 428 | 432 | 433 | 437
  3) Pain/discomfort (week 52) | 0.76 (22.31) | 2.52 (22.04) | 3.15 (23.29) | 2.12 (21.73)
  3) Pain/discomfort (week 78): number analyzed (Participants) | 425 | 425 | 427 | 441
  3) Pain/discomfort (week 78) | 3.06 (20.39) | 2.35 (22.66) | 4.07 (22.28) | 3.63 (22.38)
  4) Psychosocial (week 26): number analyzed (Participants) | 438 | 437 | 437 | 447
  4) Psychosocial (week 26) | 2.69 (13.32) | 4.30 (15.05) | 2.98 (14.86) | 2.10 (13.21)
  4) Psychosocial (week 52): number analyzed (Participants) | 428 | 432 | 434 | 437
  4) Psychosocial (week 52) | 3.12 (14.55) | 5.19 (15.04) | 3.97 (16.46) | 2.53 (14.09)
  4) Psychosocial (week 78): number analyzed (Participants) | 424 | 425 | 427 | 440
  4) Psychosocial (week 78) | 3.83 (14.89) | 5.36 (15.62) | 3.73 (16.22) | 3.29 (14.53)
  IWQOL-Lite-CT Total (week 26): number analyzed (Participants) | 438 | 437 | 437 | 447
  IWQOL-Lite-CT Total (week 26) | 2.88 (12.11) | 3.62 (13.37) | 2.95 (13.87) | 2.05 (12.05)
  IWQOL-Lite-CT Total (week 52): number analyzed (Participants) | 428 | 432 | 433 | 437
  IWQOL-Lite-CT Total (week 52) | 2.67 (13.01) | 4.43 (13.59) | 3.64 (15.22) | 2.17 (12.86)
  IWQOL-Lite-CT Total (week 78): number analyzed (Participants) | 424 | 425 | 427 | 440
  IWQOL-Lite-CT Total (week 78) | 3.45 (13.32) | 4.73 (14.07) | 3.77 (14.97) | 3.16 (13.76)

43. Secondary Outcome: Change in CoEQ: Scores From the 4 Domains and the 19 Items
Description: Change from baseline (week 0) in Control of Eating Questionnaire (CoEQ) was evaluated at weeks (wk) 26, 52 and 78. The CoEQ comprised 19 items to assess the intensity and type of food cravings, as well as subjective sensation of appetite and mood, with the 4 domains: 'craving control' (items 9-12, 19), 'positive mood' (items 5-8), 'craving for savoury' (items 4, 16-18) and 'craving for sweet' (items 3, 13-15). The 19 items were scored on an 11-point graded response scale ranging from 10 to 0, with items relating to each of the 4 domains being averaged to create a final score. A low score in the domains 'craving for sweet and 'craving for savoury' represents a low level of craving; whereas a high score in the domains 'craving control' and 'positive mood' represents good control and a good mood, respectively. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 26, week 52, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 466 | 465 | 465 | 467
Score on a scale
  1) Feeling of hunger (wk 26): number analyzed (Participants) | 438 | 435 | 437 | 446
  1) Feeling of hunger (wk 26) | -0.41 (2.61) | -0.37 (2.58) | -0.54 (2.58) | -0.18 (2.49)
  1) Feeling of hunger (wk 52): number analyzed (Participants) | 428 | 431 | 434 | 435
  1) Feeling of hunger (wk 52) | -0.28 (2.50) | -0.23 (2.69) | -0.35 (2.65) | -0.25 (2.39)
  1) Feeling of hunger (wk 78): number analyzed (Participants) | 424 | 423 | 427 | 440
  1) Feeling of hunger (wk 78) | -0.31 (2.56) | -0.22 (2.73) | -0.36 (2.52) | -0.22 (2.55)
  2) Feeling of fullness (wk 26): number analyzed (Participants) | 438 | 435 | 436 | 446
  2) Feeling of fullness (wk 26) | -0.08 (2.66) | -0.08 (2.77) | 0.15 (2.66) | 0.15 (2.45)
  2) Feeling of fullness (wk 52): number analyzed (Participants) | 428 | 431 | 433 | 435
  2) Feeling of fullness (wk 52) | -0.02 (2.61) | -0.07 (2.64) | 0.22 (2.68) | 0.27 (2.67)
  2) Feeling of fullness (wk 78): number analyzed (Participants) | 425 | 423 | 426 | 440
  2) Feeling of fullness (wk 78) | -0.03 (2.59) | -0.09 (2.71) | 0.09 (2.74) | 0.26 (2.59)
  3) Desire to eat sweet foods (wk 26): number analyzed (Participants) | 438 | 435 | 437 | 447
  3) Desire to eat sweet foods (wk 26) | -0.41 (2.55) | -0.54 (3.02) | -0.47 (2.98) | -0.33 (2.92)
  3) Desire to eat sweet foods (wk 52): number analyzed (Participants) | 428 | 431 | 434 | 435
  3) Desire to eat sweet foods (wk 52) | -0.31 (2.74) | -0.31 (2.97) | -0.31 (3.02) | -0.45 (2.75)
  3) Desire to eat sweet foods (wk 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  3) Desire to eat sweet foods (wk 78) | -0.38 (2.51) | -0.42 (3.02) | -0.45 (2.97) | -0.49 (2.84)
  4) Desire to eat savoury foods (wk 26): number analyzed (Participants) | 438 | 434 | 437 | 447
  4) Desire to eat savoury foods (wk 26) | -0.27 (2.48) | -0.16 (2.88) | -0.30 (3.03) | -0.35 (2.74)
  4) Desire to eat savoury foods (wk 52): number analyzed (Participants) | 428 | 431 | 434 | 436
  4) Desire to eat savoury foods (wk 52) | -0.27 (2.78) | -0.21 (2.80) | -0.44 (2.94) | -0.33 (2.70)
  4) Desire to eat savoury foods (wk 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  4) Desire to eat savoury foods (wk 78) | -0.39 (2.64) | -0.39 (2.95) | -0.39 (2.80) | -0.42 (2.81)
  5) Feeling of happiness (wk 26): number analyzed (Participants) | 438 | 434 | 435 | 446
  5) Feeling of happiness (wk 26) | 0.01 (2.22) | 0.03 (2.11) | 0.04 (2.22) | 0.13 (2.21)
  5) Feeling of happiness (wk 52): number analyzed (Participants) | 428 | 431 | 433 | 435
  5) Feeling of happiness (wk 52) | 0.09 (2.25) | 0.04 (2.21) | 0.09 (2.15) | 0.14 (2.16)
  5) Feeling of happiness (wk 78): number analyzed (Participants) | 425 | 424 | 426 | 441
  5) Feeling of happiness (wk 78) | -0.05 (2.32) | -0.08 (2.21) | 0.04 (2.27) | 0.02 (2.47)
  6) Feeling of anxiousness (wk 26): number analyzed (Participants) | 437 | 435 | 437 | 444
  6) Feeling of anxiousness (wk 26) | 0.02 (2.86) | -0.18 (2.96) | 0.20 (3.22) | -0.21 (2.96)
  6) Feeling of anxiousness (wk 52): number analyzed (Participants) | 428 | 430 | 434 | 436
  6) Feeling of anxiousness (wk 52) | -0.05 (2.59) | -0.16 (2.97) | -0.06 (3.02) | 0.17 (3.14)
  6) Feeling of anxiousness (wk 78): number analyzed (Participants) | 424 | 423 | 427 | 441
  6) Feeling of anxiousness (wk 78) | 0.05 (2.69) | 0.12 (3.22) | -0.12 (2.88) | -0.01 (3.21)
  7) Feeling of alertness (wk 26): number analyzed (Participants) | 437 | 435 | 437 | 445
  7) Feeling of alertness (wk 26) | 0.11 (2.44) | 0.03 (2.61) | -0.06 (2.49) | 0.05 (2.51)
  7) Feeling of alertness (wk 52): number analyzed (Participants) | 428 | 431 | 434 | 435
  7) Feeling of alertness (wk 52) | 0.01 (2.52) | -0.14 (2.87) | -0.05 (2.50) | -0.05 (2.56)
  7) Feeling of alertness (wk 78): number analyzed (Participants) | 423 | 424 | 426 | 441
  7) Feeling of alertness (wk 78) | 0.10 (2.43) | -0.04 (2.69) | 0.04 (2.48) | -0.01 (2.64)
  8) Feeling of contentment (wk 26): number analyzed (Participants) | 438 | 435 | 437 | 447
  8) Feeling of contentment (wk 26) | 0.05 (2.37) | 0.04 (2.38) | 0.18 (2.37) | 0.18 (2.14)
  8) Feeling of contentment (wk 52): number analyzed (Participants) | 428 | 431 | 434 | 436
  8) Feeling of contentment (wk 52) | 0.04 (2.35) | 0.08 (2.48) | 0.13 (2.40) | 0.20 (2.29)
  8) Feeling of contentment (wk 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  8) Feeling of contentment (wk 78) | -0.04 (2.50) | -0.03 (2.41) | 0.17 (2.38) | 0.17 (2.39)
  9) Food cravings during last 7 days (wk 26): number analyzed (Participants) | 437 | 433 | 437 | 445
  9) Food cravings during last 7 days (wk 26) | -0.59 (2.87) | -0.41 (2.94) | -0.37 (2.69) | -0.46 (2.85)
  9) Food cravings during last 7 days (wk 52): number analyzed (Participants) | 428 | 431 | 433 | 435
  9) Food cravings during last 7 days (wk 52) | -0.40 (2.99) | -0.30 (2.96) | -0.25 (2.86) | -0.21 (3.09)
  9) Food cravings during last 7 days (wk 78): number analyzed (Participants) | 423 | 423 | 427 | 441
  9) Food cravings during last 7 days (wk 78) | -0.47 (2.87) | -0.28 (2.90) | -0.38 (2.91) | -0.33 (3.05)
  10) Strength of food cravings (wk 26): number analyzed (Participants) | 438 | 436 | 436 | 447
  10) Strength of food cravings (wk 26) | -0.50 (2.75) | -0.33 (2.93) | -0.25 (2.79) | -0.35 (2.77)
  10) Strength of food cravings (wk 52): number analyzed (Participants) | 428 | 432 | 434 | 436
  10) Strength of food cravings (wk 52) | -0.23 (2.84) | -0.14 (2.90) | -0.21 (2.74) | -0.30 (2.77)
  10) Strength of food cravings (wk 78): number analyzed (Participants) | 425 | 425 | 427 | 439
  10) Strength of food cravings (wk 78) | -0.20 (2.89) | -0.28 (2.99) | -0.32 (2.85) | -0.38 (2.79)
  11) Difficulty to resist food cravings (wk 26): number analyzed (Participants) | 438 | 436 | 437 | 446
  11) Difficulty to resist food cravings (wk 26) | -0.46 (2.74) | -0.38 (3.02) | -0.46 (3.04) | -0.17 (2.84)
  11) Difficulty to resist food cravings (wk 52): number analyzed (Participants) | 428 | 431 | 434 | 436
  11) Difficulty to resist food cravings (wk 52) | 0.00 (2.79) | -0.23 (3.04) | -0.42 (3.16) | -0.26 (3.04)
  11) Difficulty to resist food cravings (wk 78): number analyzed (Participants) | 424 | 424 | 427 | 441
  11) Difficulty to resist food cravings (wk 78) | -0.04 (3.02) | -0.32 (3.20) | -0.24 (3.14) | -0.22 (2.96)
  12) Eating in response to food cravings (wk 26): number analyzed (Participants) | 438 | 436 | 437 | 446
  12) Eating in response to food cravings (wk 26) | -0.40 (2.49) | -0.15 (2.78) | -0.17 (2.78) | -0.27 (2.64)
  12) Eating in response to food cravings (wk 52): number analyzed (Participants) | 428 | 432 | 434 | 435
  12) Eating in response to food cravings (wk 52) | -0.04 (2.55) | -0.11 (2.85) | -0.25 (2.73) | -0.17 (2.75)
  12) Eating in response to food cravings (wk 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  12) Eating in response to food cravings (wk 78) | -0.02 (2.67) | 0.01 (2.76) | -0.17 (2.96) | -0.25 (2.73)
  13) Cravings for chocolate (wk 26): number analyzed (Participants) | 437 | 437 | 436 | 447
  13) Cravings for chocolate (wk 26) | -0.27 (2.69) | -0.03 (2.93) | -0.14 (2.94) | -0.15 (2.78)
  13) Cravings for chocolate (wk 52): number analyzed (Participants) | 427 | 431 | 434 | 435
  13) Cravings for chocolate (wk 52) | -0.28 (2.58) | 0.03 (2.93) | 0.06 (2.87) | 0.03 (2.85)
  13) Cravings for chocolate (wk 78): number analyzed (Participants) | 425 | 424 | 426 | 440
  13) Cravings for chocolate (wk 78) | -0.08 (2.74) | 0.00 (2.87) | 0.06 (3.01) | 0.06 (3.04)
  14) Cravings for other sweet foods (wk 26): number analyzed (Participants) | 437 | 436 | 437 | 447
  14) Cravings for other sweet foods (wk 26) | -0.33 (2.65) | -0.31 (2.91) | -0.36 (2.82) | -0.33 (2.82)
  14) Cravings for other sweet foods (wk 52): number analyzed (Participants) | 428 | 432 | 434 | 436
  14) Cravings for other sweet foods (wk 52) | -0.33 (2.79) | -0.34 (2.93) | -0.31 (2.96) | -0.09 (2.90)
  14) Cravings for other sweet foods (wk 78): number analyzed (Participants) | 425 | 425 | 427 | 441
  14) Cravings for other sweet foods (wk 78) | -0.20 (2.84) | -0.14 (3.01) | -0.40 (2.93) | -0.22 (2.87)
  15) Cravings for fruit or fruit juice (wk 26): number analyzed (Participants) | 437 | 437 | 436 | 446
  15) Cravings for fruit or fruit juice (wk 26) | -0.20 (3.05) | -0.03 (3.27) | -0.09 (3.04) | -0.07 (3.09)
  15) Cravings for fruit or fruit juice (wk 52): number analyzed (Participants) | 428 | 431 | 432 | 433
  15) Cravings for fruit or fruit juice (wk 52) | -0.40 (2.99) | -0.01 (3.34) | -0.22 (3.07) | -0.08 (3.02)
  15) Cravings for fruit or fruit juice (wk 78): number analyzed (Participants) | 425 | 425 | 426 | 439
  15) Cravings for fruit or fruit juice (wk 78) | -0.14 (2.97) | -0.11 (3.51) | -0.02 (3.12) | -0.33 (2.88)
  16) Cravings for dairy foods (wk 26): number analyzed (Participants) | 437 | 437 | 437 | 447
  16) Cravings for dairy foods (wk 26) | -0.23 (3.06) | -0.20 (2.90) | -0.37 (3.02) | -0.27 (2.83)
  16) Cravings for dairy foods (wk 52): number analyzed (Participants) | 427 | 430 | 434 | 435
  16) Cravings for dairy foods (wk 52) | -0.42 (2.96) | -0.30 (2.97) | -0.41 (2.86) | 0.04 (2.89)
  16) Cravings for dairy foods (wk 78): number analyzed (Participants) | 425 | 425 | 426 | 439
  16) Cravings for dairy foods (wk 78) | -0.30 (3.00) | -0.20 (2.95) | -0.45 (2.86) | -0.20 (2.81)
  17) Cravings for starchy foods (wk 26): number analyzed (Participants) | 436 | 436 | 436 | 447
  17) Cravings for starchy foods (wk 26) | -0.42 (2.65) | -0.24 (2.56) | -0.49 (2.75) | -0.42 (2.86)
  17) Cravings for starchy foods (wk 52): number analyzed (Participants) | 426 | 430 | 434 | 435
  17) Cravings for starchy foods (wk 52) | -0.54 (2.86) | -0.35 (2.68) | -0.62 (2.80) | -0.28 (2.68)
  17) Cravings for starchy foods (wk 78): number analyzed (Participants) | 423 | 423 | 426 | 441
  17) Cravings for starchy foods (wk 78) | -0.44 (2.94) | -0.32 (2.76) | -0.61 (2.86) | -0.36 (2.72)
  18) Cravings for savoury foods (wk 26): number analyzed (Participants) | 437 | 437 | 437 | 443
  18) Cravings for savoury foods (wk 26) | -0.41 (2.74) | -0.16 (2.69) | -0.49 (2.85) | -0.40 (2.70)
  18) Cravings for savoury foods (wk 52): number analyzed (Participants) | 427 | 431 | 434 | 436
  18) Cravings for savoury foods (wk 52) | -0.41 (2.85) | -0.20 (2.82) | -0.56 (2.72) | -0.37 (2.73)
  18) Cravings for savoury foods (wk 78): number analyzed (Participants) | 423 | 422 | 427 | 440
  18) Cravings for savoury foods (wk 78) | -0.27 (2.88) | -0.16 (2.87) | -0.48 (2.95) | -0.34 (2.60)
  19) Difficulty to control eating in general(wk 26): number analyzed (Participants) | 436 | 437 | 437 | 447
  19) Difficulty to control eating in general(wk 26) | -0.47 (2.68) | -0.69 (2.77) | -0.49 (2.69) | -0.51 (2.70)
  19) Difficulty to control eating in general(wk 52): number analyzed (Participants) | 428 | 432 | 434 | 436
  19) Difficulty to control eating in general(wk 52) | -0.32 (2.76) | -0.59 (2.86) | -0.56 (2.75) | -0.51 (2.73)
  19) Difficulty to control eating in general(wk 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  19) Difficulty to control eating in general(wk 78) | -0.40 (2.71) | -0.59 (2.88) | -0.54 (2.71) | -0.51 (2.81)
  Craving control: items 9-12, 19 (wk 26): number analyzed (Participants) | 438 | 437 | 437 | 447
  Craving control: items 9-12, 19 (wk 26) | 0.49 (2.13) | 0.39 (2.18) | 0.35 (2.16) | 0.35 (2.10)
  Craving control: items 9-12, 19 (wk 52): number analyzed (Participants) | 428 | 432 | 434 | 436
  Craving control: items 9-12, 19 (wk 52) | 0.20 (2.20) | 0.27 (2.26) | 0.34 (2.21) | 0.29 (2.18)
  Craving control: items 9-12, 19 (wk 78): number analyzed (Participants) | 425 | 425 | 427 | 441
  Craving control: items 9-12, 19 (wk 78) | 0.22 (2.30) | 0.29 (2.35) | 0.33 (2.29) | 0.34 (2.19)
  Positive mood: items 5-8 (wk 26): number analyzed (Participants) | 438 | 435 | 437 | 447
  Positive mood: items 5-8 (wk 26) | 0.04 (1.51) | 0.07 (1.43) | -0.01 (1.61) | 0.15 (1.47)
  Positive mood: items 5-8 (wk 52): number analyzed (Participants) | 428 | 431 | 434 | 436
  Positive mood: items 5-8 (wk 52) | 0.04 (1.50) | 0.03 (1.54) | 0.05 (1.60) | 0.03 (1.57)
  Positive mood: items 5-8 (wk 78): number analyzed (Participants) | 425 | 424 | 427 | 441
  Positive mood: items 5-8 (wk 78) | -0.01 (1.57) | -0.07 (1.52) | 0.09 (1.55) | 0.05 (1.74)
  Craving for savoury: items 4, 16-18 (wk 26): number analyzed (Participants) | 437 | 437 | 437 | 447
  Craving for savoury: items 4, 16-18 (wk 26) | -0.33 (1.88) | -0.19 (1.94) | -0.41 (2.07) | -0.36 (1.89)
  Craving for savoury: items 4, 16-18 (wk 52): number analyzed (Participants) | 428 | 432 | 434 | 436
  Craving for savoury: items 4, 16-18 (wk 52) | -0.41 (2.01) | -0.27 (1.95) | -0.51 (2.11) | -0.24 (1.88)
  Craving for savoury: items 4, 16-18 (wk 78): number analyzed (Participants) | 425 | 425 | 427 | 441
  Craving for savoury: items 4, 16-18 (wk 78) | -0.35 (2.06) | -0.26 (2.12) | -0.48 (2.08) | -0.33 (1.93)
  Craving for sweet: items 3, 13-15 (wk 26): number analyzed (Participants) | 437 | 437 | 437 | 447
  Craving for sweet: items 3, 13-15 (wk 26) | -0.30 (1.88) | -0.23 (2.12) | -0.26 (2.10) | -0.22 (2.01)
  Craving for sweet: items 3, 13-15 (wk 52): number analyzed (Participants) | 428 | 432 | 434 | 436
  Craving for sweet: items 3, 13-15 (wk 52) | -0.33 (1.97) | -0.15 (2.17) | -0.19 (2.19) | -0.15 (2.06)
  Craving for sweet: items 3, 13-15 (wk 78): number analyzed (Participants) | 425 | 425 | 427 | 441
  Craving for sweet: items 3, 13-15 (wk 78) | -0.20 (1.94) | -0.16 (2.22) | -0.20 (2.20) | -0.24 (2.06)

ADVERSE EVENTS:
Time Frame: Week 0 to week 83 (78 weeks treatment period + 5 weeks follow-up period). Results are based on the safety analysis set (SAS), which comprised all randomised participants who received at least one dose of trial product.
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
All-Cause Mortality (participants affected / at risk) | 5/466 | 4/464 | 1/465 | 3/466
Serious Adverse Events (participants affected / at risk) | 64/466 | 47/464 | 44/465 | 58/466
Other Adverse Events (participants affected / at risk) | 222/466 | 234/464 | 232/465 | 239/466
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=466) | Oral Semaglutide 7 mg (N=464) | Oral Semaglutide 14 mg (N=465) | Sitagliptin 100 mg (N=466)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 4 (4)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract diabetic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exostosis of external ear canal (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Laparoscopic surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 4 (4)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyp (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy proliferative (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Septic phlebitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=466) | Oral Semaglutide 7 mg (N=464) | Oral Semaglutide 14 mg (N=465) | Sitagliptin 100 mg (N=466)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (29) | 13 (17) | 20 (25) | 29 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (35) | 25 (31) | 24 (25) | 29 (35)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 14 (15) | 32 (32) | 14 (15)
Diabetic retinopathy (Eye disorders) | 27 (27) | 24 (25) | 16 (16) | 26 (27)
Diarrhoea (Gastrointestinal disorders) | 44 (62) | 53 (81) | 56 (74) | 37 (44)
Headache (Nervous system disorders) | 29 (37) | 30 (40) | 36 (50) | 36 (57)
Hypertension (Vascular disorders) | 29 (32) | 24 (27) | 26 (26) | 29 (29)
Influenza (Infections and infestations) | 29 (35) | 24 (28) | 18 (21) | 30 (35)
Nasopharyngitis (Infections and infestations) | 53 (74) | 49 (65) | 47 (57) | 47 (69)
Nausea (Gastrointestinal disorders) | 34 (42) | 62 (74) | 70 (88) | 31 (39)
Upper respiratory tract infection (Infections and infestations) | 36 (53) | 35 (50) | 26 (34) | 32 (49)
Urinary tract infection (Infections and infestations) | 29 (32) | 21 (26) | 23 (30) | 26 (32)
Vomiting (Gastrointestinal disorders) | 13 (15) | 27 (41) | 42 (82) | 19 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT02607865/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT02607865/SAP_001.pdf